CLINICAL TRIAL: NCT07049692
Title: Evaluation of the Efficacy and Safety of Hyperbaric Oxygen in Patients After Endovascular Treatment for Acute Ischemic Stroke: A Multicenter, Open-label, Randomized Controlled Clinical Trial
Brief Title: Hyperbaric Oxygen After Stroke Thrombectomy: A Multicenter Randomized Trial on Safety and Efficacy
Acronym: NOTICE-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Jing Yang, Hyperbaric Oxygen Department, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-KE-357-2; 2025-3-4-2 (Registry Identifier: NOTICE-1)
Record Dates: First submitted 2025-06-13; First posted 2025-07-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-10

CONDITIONS: Acute Ischemic Stroke
Keywords: HBO; acute ischemic stroke; endovascular treatment
MeSH Terms: conditions — Ischemic Stroke | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperbaric oxygen therapy (Experimental)
  Interventions: Other: Hyperbaric Oxygen Therapy
- Control group (Other)
  Interventions: Other: Conventional therapy group

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — 1.6 atmosphere absolute (1.6 ATA), HBO treatment administrated via mask or hood, one 60 minutes session, once daily, 5 days a week (can be non consecutive days), with a total of 10 sessions.
  Arms: hyperbaric oxygen therapy
Other: Conventional therapy group — Conventional therapy
  Arms: Control group

SUMMARY:
1. The goal of this clinical trial is to evaluate the efficacy and safety of hyperbaric oxygen (HBO)in stroke patients after endovascular treatment
2. The main questions it aims to answer is:

   Whether HBO can improve the prognosis of ischemic stroke patients after endovascular treatment?
3. Participants will:

receive HBO (1.6 Atmosphere Absolute，1.6ATA)，Once a day, for 1 hour each time, for 5 days a week (it can be non-consecutive days), the total course of treatment is 10 times.

undergo three scheduled face to face or telephone follow-up assessments during the 12-month period following HBO.

ELIGIBILITY:
Inclusion Criteria:

* 35-75 years
* The symptoms and signs are consistent with acute anterior circulation ischemic stroke. The immediate postoperative angiographic recanalization grade was ≥ 2b.
* Neurological deficit score at the time of enrollment: 5 ≤ NIHSS ≤ 15 points
* Consciousness status (NIHSS 1a-1b items): 0-1 point
* Pre-stroke functional status (mRS score): 0-1
* Time from surgery to randomization grouping: ≤ 72 hours
* Patient or legal representative who signed the informed consent form
* Preoperative CT angiography or magnetic resonance angiography confirmed large vessel occlusion (internal carotid artery or middle cerebral artery M1 segment) that was consistent with the symptoms and signs; And the area supplied by the middle cerebral artery in the brain is less than 1/3.
* A lberta S troke P rogram E arly C T S core ≥ 6

Exclusion Criteria:

* Subjects with HBO contraindications or intolerance
* Postprocedural imaging identified either procedure-related subarachnoid hemorrhage or hemorrhagic transformation
* Based on the medical history, it is suspected that the cerebral embolism is caused by sepsis or infective endocarditis
* Expected lifespan < 90 days
* Severe heart, liver and kidneys failure
* Pregnancy
* Hereditary or acquired bleeding tendency, deficiency of coagulation factors, recent use of oral anticoagulants with an international normalized ratio (INR) > 3 or activated partial thromboplastin time (APTT) exceeding the normal value by more than 3 times
* Baseline platelet count < 50×10 9/L
* Baseline blood glucose is less than 2.78 mmol/L or greater than 22.2 mmol/L.
* Unstable vital signs (heart rate ≤ 50 beats/min or ≥ 120 beats/min, oxygen saturation ≤ 90%, respiration ≥ 30 breaths/min or ≤ 10 breaths/min);
* Hypertension that cannot be controlled by medication: Systolic blood pressure ≥ 160 mmHg, or diastolic blood pressure ≥ 100 mmHg;
* Suspected of having acute myocardial infarction;
* Currently involving in the research of other projects related to drugs or medical devices.
* CT or MRI scans revealed intracranial tumors (except for cerebellar meningiomas) and intracranial arteriovenous malformations.
* Based on the medical history and CT or MRI findings, a diagnosis of internal carotid artery dissection or aortic dissection is suspected;
* Based on the medical history and CT or MRI findings, cerebral vasculitis is suspected.
* Based on the clinical evidence of multiple vascular regions being occluded (either in the bilateral anterior circulation or anterior/posterior circulation) or bilateral infarction or multi-region infarction as detected by CT angiography or magnetic resonance angiography;
* CT or magnetic resonance imaging shows a significant midline shift effect (> 0.5 cm);
* CT angiography or magnetic resonance angiography confirmed the presence of cerebral vasculitis or cerebral vasculitis syndrome;

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a favorable prognosis (mRS score of 0-2 ) after randomization at 90 (±7) days | Day 90 (±7) post-randomization
  Modified Rankin Scale (mRS) is defined as the gold standard for measuring global functional outcomes after stroke: 0-1 indicating functional independence, 0-2 favorable prognosis, defining functional independence, 4-5 Severely disabled, 6 death. Higher mRS scores indicate worse prognosis.

SECONDARY OUTCOMES:
Core infarction volume on Diffusion-Weighted Imaging | Day 10 (±1）post-randomization
  The effectiveness of HBO for patients with acute ischemic stroke was evaluated based on the core cerebral infarction volume.
National Institutes of Health Stroke Scale (NIHSS）score [(0, Normal)-(42, worst)] | Day 10(±1) NIHSS score post-randomization
  The effectiveness of HBO therapy in patients with acute ischemic stroke undergoing endovascular treatment was evaluated based on the improvement rate of NIHSS score day 10 post-randomization.
mRS score [ (0, Normal)-(6, worst)] | Day 10 (±1）post-randomization; Day 30(±3) post-randomization; Day 180(±14) post-randomization; Day 360(±30) post-randomization.
  To assess the effectiveness of HBO treament for ischemic stroke using mRS score on day 10, 30, 90 and 360 post-randomization
Distribution of mRS score [(0, normal)-6(worst)] | Day 90 (±7) post-randomization
  mRS (0-1): the proportion of functional independence; mRS (0-2): the proportion of good prognosis; mRS (4-6) : the proportion of severe disability.
Bartherl index (BI)[(0, worst)-(100, normal)] | Day 30(±3), 90(±7) , 180(±14) and 360 (±30) post-randomization
  Functional independence was assessed using the BI
EuroQol 5-Dimensions(EQ-5D)[(0, worst)-(100, normal)] | Day 30(±3), 90(±7), 180(±14), 360(±30) post-randomization
  Health-related quality of life was measured using EQ-5D.
Stroke recurrence rate | Day 30(±3) , 90(±7d), 180(±14d) and 360(±30) post-randomization
  New symptoms persisting for > 24 hours and new lension on the DWI.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
1. Primary/secondary efficacy endpoint data
  2. Safety data
  3. Baseline characteristic dataset
  4. Plan Deviation Record
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 31/12/2028-31/12/2043
Access Criteria: Qualified researchers can access de-identified IPD, protocols, and analysis plans through [Repository Name] after submitting a research proposal and signing a Data Use Agreement. Data is available in CDISC formats for non-commercial research only, with results required within 24 months. Re-identification and commercial use are prohibited.